CLINICAL TRIAL: NCT06596070
Title: Clinical Study of Intestinal Barrier Dysfunction in Patients After Gastrointestinal Surgery
Brief Title: Clinical Study of Intestinal Barrier Dysfunction After Gastrointestinal Surgery
Status: Not yet recruiting | Type: Observational
Sponsor: The Second Affiliated Hospital of Kunming Medical University (Other)
Responsible Party: Principal Investigator, Weiming Li, Investigator, The Second Affiliated Hospital of Kunming Medical University
Other Study IDs: PJ-2024-124
Record Dates: First submitted 2024-09-07; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Intestinal Barrier Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Intestinal barrier dysfunction group
  Interventions: Other: No intervention was carried out
- Non-intestinal barrier dysfunction group
  Interventions: Other: No intervention was carried out

INTERVENTIONS:
Other: No intervention was carried out — This study is an observational study and no intervention was performed on the patients.

SUMMARY:
The goal of this observational study is to explore the clinical influences associated with the development of intestinal barrier dysfunction in patients undergoing gastrointestinal surgery. The main question it aims to answer is:What clinical factors increase the probability of developing intestinal barrier dysfunction in patients after gastrointestinal surgery?

ELIGIBILITY:
Inclusion Criteria:

* men or women aged 18-80 years
* expected feasible abdominal surgical treatment (partial gastrectomy, colorectal resection)
* no preoperative intestinal barrier dysfunction
* patients voluntarily participated in this study and signed an informed consent form.

Exclusion Criteria:

* Patients or their families refused to participate in this study
* chronic inflammatory diseases (e.g. inflammatory bowel disease, chronic hepatitis, chronic pancreatitis, chronic peptic ulcer, etc.)
* history of antibiotic administration in the last 2 weeks
* severe cognitive impairment and other inability to cooperate preoperative neoadjuvant radiotherapy
* combined with severe hepatic, renal, and cardiac insufficiency patients.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People undergoing gastrointestinal surgery
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
operating time | During surgery
  Record the patient's surgical time

SECONDARY OUTCOMES:
nutritional status | Preoperative
  Patients were assessed for risk of malnutrition by the Nutritional Risk Screening Scale (NRS-2002). A score of ≥3 indicated that the patient was at risk of malnutrition.
bowel habit | Preoperative
  The patient was asked whether there were increased frequency of stool, changes in stool characteristics, constipation and other conditions before surgery
Surgical Procedures | During surgery
  Record whether the patient underwent laparoscopic surgery or open surgery
hemorrhage | During surgery
  Record the patient's intraoperative bleeding volume
Albumin | Preoperative and postoperative 24 hours
  Record the patient's albumin levels before and 24 hours after surgery
Infection indicators | Preoperative and postoperative 24 hours
  Record the values of PCT, IL-6, and CRP of patients before and 24 hours after surgery
age | Preoperative
gender | Preoperative
Body Mass Index | Preoperative
diabetes | Preoperative
  Record whether the patient has diabetes
enteral nutrition | The average observation time is 2 weeks after surgery.
  Record the start time of enteral nutrition for patients after surgery.
Exhaust and defecation time | The average observation time is one week after surgery
  Record the time of the patient's first exhaust and first bowel movement after surgery

IPD SHARING:
Plan to Share IPD: Undecided
Research not yet completed